CLINICAL TRIAL: NCT02220023
Title: Dynamic Assessment of Right Ventricular Function With Inhaled Nitric Oxide During Cardiac MRI
Acronym: iNO
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Principal Investigator, Evan Brittain, Assistant Professor, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 140068
Record Dates: First submitted 2014-08-14; First posted 2014-08-19 (Estimated); Last update posted 2017-02-13 (Actual); Status verified 2017-02

CONDITIONS: Pulmonary Vascular Disorder
MeSH Terms: interventions — Nitric Oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nitric Oxide (Experimental): 40 ppm, one time administration, inhaled.
  Interventions: Drug: INOmax Inhalation

INTERVENTIONS:
Drug: INOmax Inhalation
  Other Names: nitric oxide; NDA 20-845

SUMMARY:
The purpose of the study is to measure RV ejection fraction (RVEF), pulmonary flow, and pulmonary perfusion before and after exposure to inhaled nitric oxide in patients with pulmonary arterial hypertension (PAH) who are known to be vasodilator-responsive based on invasive catheterization as well as healthy subjects. Measurements will also be made after high flow oxygen alone to test the relative vasodilatory effect of oxygen and NO. The investigators hypothesize is that inhaled nitric oxide during cardiac MRI can be used to measure dynamic changes in RV-pulmonary vascular function in patients with vasodilator-responsive PAH.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 or older of the Vanderbilt Center for Pulmonary Vascular Disease. Vasodilator-responsive patients will be identified based on prior response to inhaled nitric oxide during invasive right heart catheterization
* Healthy subjects age 18 or older not known to have cardiopulmonary disease

Exclusion Criteria:

* Standard conventional contraindications for cardiac magnetic resonance (CMR) imaging
* Allergy or contraindication to Magnevist (gadopentetate dimeglumine) contrast
* Concurrent intravenous epoprostenol infusion in whom performance of CMR is cumbersome
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-07; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Right ventricular ejection fraction (RVEF) before and after inhaled nitric oxide exposure | At time of procedure

SECONDARY OUTCOMES:
Pulmonary flow | Baseline, after 4 minutes high flow oxygen, after 4 minutes high flow oxygen plus nitric oxide
Pulmonary perfusion | Baseline, after 4 minutes of high flow oxygen, after 4 minutes of high flow oxygen plus nitric oxide
Estimates of pulmonary vascular resistance | At Baseline, after 4 minutes of high flow oxygen, after 4 minutes of high flow oxygen plus nitric oxide
Pulmonary transit time | At baseline, after 4 minutes high flow oxygen, after 4 minutes high flow oxygen plus nitric oxide
Pulmonary artery compliance | At baseline, after 4 minutes high flow oxygen, after 4 minutes high flow oxygen plus nitric oxide

CONTACTS AND LOCATIONS:
Overall Officials: Evan L Brittain, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States